CLINICAL TRIAL: NCT03702868
Title: A Prospective Cohort Study of Relationship Between Gut Microbiome and Adjuvant Chemotherapy in Patients With Early Breast Cancer
Brief Title: Relationship Between Gut Microbiome and Adjuvant Chemotherapy in Patients With Early Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Difficulty accruing subjects the study accrual was closed
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Professor Zhongyu Yuan, Sun Yat-sen University
Other Study IDs: SYSUCC-011
Record Dates: First submitted 2018-09-02; First posted 2018-10-11 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Adjuvant Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fresh fecal sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Breast cancer is the most common cause of cancer death in women. Adjuvant chemotherapy significantly reduces the risk of recurrence of high-risk breast cancer. However, about 30% of patients still have distant metastasis or local recurrence after chemotherapy. Moreover, 60% of patients had 3-4 degrees of adverse drug reactions during chemotherapy.

The purpose of the study is to investigate relationship between gut microbiome and adjuvant chemotherapy in early breast cancer patients.

DETAILED DESCRIPTION:
Breast cancer is the most common cause of cancer death in women. Adjuvant chemotherapy significantly reduces the risk of recurrence of high-risk breast cancer. However, about 30% of patients still have distant metastasis or local recurrence after chemotherapy. Moreover, 60% of patients had 3-4 degrees of adverse drug reactions during chemotherapy.

The human gut microbiota have been considered the most important microecosystem living in symbiosis with the body. It is identified as a crucial determinant in cancer occurrence and development . Besides, Gut microbial alterations may influence the therapy efficacy and adverse drug event.

We collect the fresh tail stool sample 24h before adjuvant chemotherapy and 24h after adjuvant chemotherapy then the composition of intestinal microbiota and subsequent short-term alterations are analysed by 16srRNA sequencing.The purpose of the study is to investigate relationship between gut microbiome and adjuvant chemotherapy in early breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically diagnosed stage I-III breast cancer;
* Plan to receive adjuvant chemotherapy in our hospital;
* Sign the informed consent;
* Good compliance and willing to follow up.

Exclusion Criteria:

* Those who have started receiving adjuvant chemotherapy;
* Chemotherapy contraindications;

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: early breast cancer patients ready to receive adjuvant chemotherapy.
Sampling Method: Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
The incidence of chemotherapy related adverse reaction | 1 years
  chemotherapy related adverse reaction are assessed by CTCAE protocol

SECONDARY OUTCOMES:
disease free survival | 5years
  the length of time after surgery during which no breast cancer is found

CONTACTS AND LOCATIONS:
Overall Officials: Zhong-yu Yuan, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided